CLINICAL TRIAL: NCT04309045
Title: Assessment of Cost-effectiveness in Two Empirically-based Psychotherapies for Borderline Personality Disorder: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Yuval Bloch, Professor, Shalvata Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0011-19-SHA
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Treatment 1:Dialectical Behavior Therapy (DBT); Treatment 2:Dynamic Deconstructive Psychotherapy (DDP); Placebo
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DBT (Experimental): Standard DBT treatment
  Interventions: Behavioral: DBT
- DDP (Active Comparator): dynamic deconstructive psychotherapy (DDP) treatment, is part of a trend of dynamic therapies to treat borderline personality disorder. DDP is a treatment specifically developed for a population with more severe symptoms those dealing with borderline personality disorder.
  Interventions: Behavioral: DDP
- control group (Placebo Comparator): patients on the waiting list for treatment, or patients in the hospital under routine care. Which will form the control group.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: DBT — Today, the most well-known and established treatment for borderline personality disorder is Dialectical Behavior Therapy (DBT) that developed by Marsha Linhan in the 1990s. DBT is currently used in other disorders such as: eating disorders, addictions, impulse control problems and bipolar disorder. Various studies have found a beneficial effect for this treatment in various areas: decreased suicidal thoughts and attempts and self-harm behaviors, improvements in suicide attempts, anger levels, impulsive behaviors, depressive symptoms, The use of drugs, the percentage of dropouts from treatment, number Hospitalization and general function.
  Arms: DBT
Behavioral: DDP — DDP treatment is part of a trend of dynamic therapies to treat borderline personality disorder. The DDP focuses on deficiencies in the emotional experience processing and is performed in the form of weekly, individual sessions with a trained therapist over a 12-18 month period. Treatment is based on the need to correct three neurocognitive functions responsible for adaptive processing of emotional experiences: association (the ability to recognize, understand their existence, and experience a sequence of emotional experiences), attribution (the ability to make complex attributions about the self and others), and the ability to make realistic attribution, about the self and the other. Interventions that activate these three functions are the basis for DDP treatment.
  Arms: DDP
Other: control group — Patients on the waiting list for treatment, or patients in the hospital under routine care.
  Arms: control group

SUMMARY:
Patients suffering from borderline personality disorder (BPD) are considered frequent utilizers of psychiatric emergency rooms and of psychiatric hospitalizations. Nonetheless, recent studies challenge the effectiveness of psychiatric hospitalizations in reducing BPD symptoms, and some have even indicated potentially harmful effects such as increasing suicide risk post-discharge. These findings highlight the importance of effective outpatient treatments for BPD patients in public psychiatric hospital settings. In this study we aim to assess the effectiveness and cost-effectiveness of two empirically-based treatments for BPD: dialectical behavior therapy (DBT) and dynamic deconstructive psychotherapy (DDP).

DETAILED DESCRIPTION:
In this study we aim to assess the effectiveness and cost-effectiveness of two empirically-based treatments for BPD: dialectical behavior therapy (DBT) and dynamic deconstructive psychotherapy (DDP). Sixty-eight participants with BPD will be randomized to each of two treatment groups. Participants and therapists will be recruited from the Shalvata MHC, a 139-bed psychiatric institution with outpatient units serving a population of more than 600,000 people in Israel. A blinded research assistant will administer primary and secondary outcome measures every 3 months during the 12 months of treatment and at the end of the 6-month naturalistic follow-up period after ending treatment with DDP or DBT. Therapist adherence will be systematically assessed in both treatments for 10% of sessions. Primary outcome measure will be comprised of the Incremental cost-effectiveness ratio (ICER), as assessed by estimating the healthcare utilization costs per incremental improvement in suicide severity. Secondary outcome measures will include BPD and depression symptom severity and quality of life. This study was submitted to the institutional review board of the Shalvata MHC in November 2019, and is expected to be approved by late Janury 2020.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 45 years old
* diagnosis of BPD,
* history of a suicide attempt within the prior year with presence of current suicidal ideation,
* agrees to participate in psychotherapy
* signed informed consent,

Exclusion Criteria:

* meet diagnostic criteria for schizophrenia, schizoaffective disorders, or have severe intellectual impairment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2024-10-22 (Estimated); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio (ICER) | The expected duration of treatment is about one year
  The measure will be assessed by comparing health care use costs in ratio to improvement on the Columbia hardware rating scale.